CLINICAL TRIAL: NCT04281004
Title: A Phase I/II Randomized, Double-Masked Placebo-Controlled Study For Determining The Safety Of Processed Amniotic Fluid (PAF) Drops After Photorefractive Keratectomy
Brief Title: Processed Amniotic Fluid (PAF) Drops After Photorefractive Keratectomy (PRK)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Mark Mifflin, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99569
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Photorefractive Keratectomy
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amniotic Fluid (AFED) (Active Comparator)
  Interventions: Biological: Amniotic Fluid (AFED)
- Saline Solution (Placebo Comparator)
  Interventions: Other: Saline Solution

INTERVENTIONS:
Biological: Amniotic Fluid (AFED) — One drop (0.25 mL) of Amniotic Fluid Eye Drops (AFED) in each eye four times daily for seven days
  Arms: Amniotic Fluid (AFED)
Other: Saline Solution — One drop (0.25 mL) of Saline Solution in each eye four times daily for seven days
  Arms: Saline Solution

SUMMARY:
This is a randomized, double-masked, placebo-controlled study to determine the safety of pAF in patients who undergo PRK.

DETAILED DESCRIPTION:
Photorefractive Keratectomy (PRK) is a common elective surgery used to correct refractive errors. We propose that amniotic fluid drops may be beneficial in promoting ocular surface healing following PRK. Purified amniotic fluid (pAF) contains anti-inflammatory, anti-microbial and regenerative factors similar to solid amniotic membrane. Individual patients will be randomized to one of two post-operative drop regimens, control eyes that will receive placebo saline solution (NaCl 0.9%, Baxter Medical), and study eyes that will receive pAF four times daily for seven days.

This is a randomized, double-masked, placebo-controlled study to determine

* the safety of pAF in patients who undergo PRK
* if pAF hastens re-epithelialization following PRK compared to placebo
* if pAF reduces post-operative pain following PRK compared to placebo
* if pAF affects visual outcome following PRK compared to placebo
* if pAF affects ocular surface staining and corneal regularity following PRK compared to placebo

ELIGIBILITY:
Inclusion:

1. Patients aged 21 years and older.
2. Patients undergoing PRK for visual correction in both eyes.
3. Willing and able to give consent for study participation and comply with study procedures, including follow-up visits.

Exclusion:

1. Patients with any active eye disease, including keratoconus or any other ectactic disorders.
2. Patients with documented uncontrolled diabetes.
3. Patients with severe dry eye as measured by corneal staining.
4. Patients with calculated PRK treatment resulting in residual stromal bed <300 um.
5. Patients who have had previous eye surgery or refractive laser procedures.
6. Patients with any active collagen vascular disease.
7. Patients who do not have potential of 20/20 or better best corrected vision in each eye.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Moran Eye Center, University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Amniotic Fluid (AFED) | Saline Solution
Started | 29; 58 eyes | 32; 64 eyes
Completed | 28; 56 eyes (One patient (two eyes) did not receive treatment due to the patient experiencing syncope during the procedure causing the procedure to be aborted.) | 32; 64 eyes
Not Completed | 1; 2 eyes | 0; 0 eyes
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: The population includes all subjects who provide informed consent and who are randomized into the trial and who have analyzable primary outcome data for at least one PRK-treated eye.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amniotic Fluid (AFED) | Saline Solution | Total
Number analyzed (Participants) | 28 | 32 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33.8 [27.6 to 38.8] | 32.7 [28.3 to 36.6] | 33.4 [28.1 to 37.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 32
  Male | 15 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 26 | 29 | 55
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 30 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 32 | 60
Current Smoker or exposed to secondhand smoke [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety - Adverse Events Including Serious Adverse Events
Description: Ocular adverse events using MedDRA and CTCAE and serious adverse events
Time Frame: Up to 12 months after the last study dose
Measure: Count of Participants; unit: Participants
Arm/Group | Amniotic Fluid (AFED) | Saline Solution
Number analyzed (Participants) | 28 | 32
Participants | 1 | 1
Statistical Analysis 1: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 1.000, Fisher Exact

2. Secondary Outcome: Time to Complete Re-epithelization
Description: Ophthalmologic assessment to determine re-epithelialization. Dimensions of the epithelial defects will be directly measured using slit lamp bio-microscopy. The baseline epithelial defect will be measured by surgeons on Day 1 at the time of surgery. A vertical and horizontal measure of defect in mm will be performed, and defect area calculated. A complete re-epithelization (absence of a defect) is defined when the measures equal zero.
Time Frame: Post-operative days 1 - 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Amniotic Fluid (AFED) | Saline Solution
Number analyzed (Participants) | 28 | 32
days | 5 (0.6) | 5 (0.5)
Statistical Analysis 1: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.869, Mixed Models Analysis; Mixed model analysis is used to account for correlation between eyes in the same participant

3. Secondary Outcome: Uncorrected Visual Acuity
Description: Ophthalmologic assessment to determine uncorrected visual acuity
Time Frame: Post-operative months 1, 3, 6, and 12
Population: Some patients missed one or more follow-up windows. We analyzed all available data.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Arm/Group | Amniotic Fluid (AFED) | Saline Solution
Number analyzed (Participants) | 27 | 31
Number analyzed (eyes) | 54 | 62
LogMAR
  Month 1 | -0.03 (0.103) | 0.04 (0.123)
  Month 3: number analyzed (Participants) | 26 | 29
  Month 3: number analyzed (eyes) | 52 | 58
  Month 3 | -0.06 (0.097) | -0.05 (0.103)
  Month 6: number analyzed (Participants) | 27 | 30
  Month 6: number analyzed (eyes) | 54 | 60
  Month 6 | -0.07 (0.085) | -0.06 (0.091)
  Month 12: number analyzed (Participants) | 25 | 26
  Month 12: number analyzed (eyes) | 50 | 51
  Month 12 | -0.09 (0.058) | -0.06 (0.107)
Statistical Analysis 1: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.007, Mixed Models Analysis — Significance of treatment effect at month 1; Mixed model analysis is used to account for correlation between eyes in the same participant
Statistical Analysis 2: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.953, Mixed Models Analysis — Significance of treatment effect at month 3; Mixed model analysis is used to account for correlation between eyes in the same participant
Statistical Analysis 3: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.841, Mixed Models Analysis — Significance of treatment effect at month 6; Mixed model analysis is used to account for correlation between eyes in the same participant
Statistical Analysis 4: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.137, Mixed Models Analysis — Significance of treatment effect at month 12; Mixed model analysis is used to account for correlation between eyes in the same participant

4. Secondary Outcome: Pain in Each Eye
Description: Patient reported pain using a visual analog scale (VAS) with 0 as no pain and 10 as worst pain
Time Frame: Post-operative days 1 - 8
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Amniotic Fluid (AFED) | Saline Solution
Number analyzed (Participants) | 28 | 32
score on a scale | 4 [2 to 7] | 5 [3 to 7]
Statistical Analysis 1: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.614, t-test, 2 sided

5. Secondary Outcome: Count of Participants Who Reported Oral Pain Medication Usage
Description: Patient reported oral pain medication usage in the first seven days of post-surgical follow-up (yes/no), where yes corresponds to any use of oral pain medication.
Time Frame: Post-operative days 1 - 8
Measure: Count of Participants; unit: Participants
Arm/Group | Amniotic Fluid (AFED) | Saline Solution
Number analyzed (Participants) | 28 | 32
Participants | 26 | 31
Statistical Analysis 1: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.594, Fisher Exact

6. Secondary Outcome: Corneal Staining in Each Eye
Description: Ocular surface staining to determine ocular dryness using an area density index with 16 index options. A0D0 equals no dry eye to A3D3 equals most severe dryness (A=area and D=density).
Time Frame: Post-operative months 1, 3, 6, and 12
Population: Subjects were analyzed for every follow-up that was collected. Some subject missed one or more follow-ups.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Amniotic Fluid (AFED) | Saline Solution
Number analyzed (Participants) | 27 | 31
Number analyzed (eyes) | 54 | 62
eyes
  Month 1: A0D0 | 33 | 42
  Month 1: A1D1 | 18 | 15
  Month 1: A1D2 | 1 | 3
  Month 1: A1D3 | 0 | 1
  Month 1: A2D2 | 2 | 1
  Month 1: A2D1 | 0 | 0
  Month 3: number analyzed (Participants) | 26 | 29
  Month 3: number analyzed (eyes) | 52 | 58
  Month 3: A0D0 | 45 | 46
  Month 3: A1D1 | 6 | 8
  Month 3: A1D2 | 0 | 2
  Month 3: A1D3 | 0 | 0
  Month 3: A2D2 | 0 | 2
  Month 3: A2D1 | 1 | 0
  Month 6: number analyzed (Participants) | 27 | 30
  Month 6: number analyzed (eyes) | 54 | 60
  Month 6: A0D0 | 46 | 52
  Month 6: A1D1 | 8 | 7
  Month 6: A1D2 | 0 | 0
  Month 6: A1D3 | 0 | 0
  Month 6: A2D2 | 0 | 1
  Month 6: A2D1 | 0 | 0
  Month 12: number analyzed (Participants) | 25 | 26
  Month 12: number analyzed (eyes) | 50 | 52
  Month 12: A0D0 | 47 | 43
  Month 12: A1D1 | 3 | 9
  Month 12: A1D2 | 0 | 0
  Month 12: A1D3 | 0 | 0
  Month 12: A2D2 | 0 | 0
  Month 12: A2D1 | 0 | 0
Statistical Analysis 1: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.663, Wilcoxon (Mann-Whitney) — Significance of treatment effect at month 1; Clustered version of the Wilcoxon test
Statistical Analysis 2: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.416, Wilcoxon (Mann-Whitney) — Significance of treatment effect at month 3; Clustered version of the Wilcoxon test
Statistical Analysis 3: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.890, Wilcoxon (Mann-Whitney) — Significance of treatment effect at month 6; Clustered version of the Wilcoxon test
Statistical Analysis 4: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.192, Wilcoxon (Mann-Whitney) — Significance of treatment effect at month 12; Clustered version of the Wilcoxon test

7. Secondary Outcome: Corneal Surface Regularity
Description: Surface Regularity Index (SRI) obtained via Zeiss Atlas 9000 Corneal Topography™. SRI is a measure of central and paracentral corneal irregularity. A lower SRI suggests more regularity of the anterior surface of the central cornea. Lower values are considered better. The minimum value is 0 and no maximum. And, a value less than 1.55 is considered normal.
Time Frame: Post-operative months 1, 3, 6, and 12
Population: Some patients missed one or more follow-up windows. We analyzed all available data.
Measure: Mean (Standard Deviation); unit: Surface regularity index
Units Other Than Participants: eyes
Arm/Group | Amniotic Fluid (AFED) | Saline Solution
Number analyzed (Participants) | 28 | 32
Number analyzed (eyes) | 56 | 64
Surface regularity index
  Month 1: number analyzed (Participants) | 24 | 30
  Month 1: number analyzed (eyes) | 48 | 60
  Month 1 | 1.34 (0.567) | 1.58 (0.748)
  Month 3: number analyzed (Participants) | 26 | 29
  Month 3: number analyzed (eyes) | 52 | 58
  Month 3 | 1.11 (0.616) | 1.07 (0.407)
  Month 6: number analyzed (Participants) | 27 | 30
  Month 6: number analyzed (eyes) | 54 | 60
  Month 6 | 1.07 (0.376) | 0.97 (0.389)
  Month 12: number analyzed (Participants) | 25 | 25
  Month 12: number analyzed (eyes) | 50 | 50
  Month 12 | 1.03 (0.459) | 1.05 (0.661)
Statistical Analysis 1: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.057, Mixed Models Analysis — Significance of treatment effect at month 1; Mixed model analysis is used to account for correlation between eyes in the same participant
Statistical Analysis 2: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.528, Mixed Models Analysis — Significance of treatment effect at month 3; Mixed model analysis is used to account for correlation between eyes in the same participant
Statistical Analysis 3: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.210, Mixed Models Analysis — Significance of treatment effect at month 6; Mixed model analysis is used to account for correlation between eyes in the same participant
Statistical Analysis 4: Comparison: Amniotic Fluid (AFED) vs Saline Solution; Test type: Superiority; p = 0.853, Mixed Models Analysis — Significance of treatment effect at month 12; Mixed model analysis is used to account for correlation between eyes in the same participant

ADVERSE EVENTS:
Time Frame: Randomization through last study visit (12 months after the last study dose), up to 56 weeks.
Description: All deaths, Serious Adverse Events, and other ocular Adverse Events regardless of seriousness were reported.
Arm/Group | Amniotic Fluid (AFED) | Saline Solution
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/32
Other Adverse Events (participants affected / at risk) | 2/28 | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amniotic Fluid (AFED) (N=28) | Saline Solution (N=32)
Intraocular pressure increased (Investigations) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The limitations of this study include small sample size and limited duration for follow-up. A larger sample size may reveal whether pAF has a protective effect against haze formation, as haze after PRK is rare. Longer duration of follow-up can reveal whether it influences final visual acuity outcomes or late haze formation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT04281004/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT04281004/SAP_003.pdf
  • Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT04281004/ICF_002.pdf